CLINICAL TRIAL: NCT03302975
Title: The Effect of a Gait Modification Training Program on Impact Loading and Running-related Injuries
Brief Title: Running Retraining to Minimize Braking Forces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Fortius Sport & Health (Other)
Responsible Party: Principal Investigator, Michael Hunt, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H16-00413
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Athletic Injuries
Keywords: Running; Biomechanics; Kinetics
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Real time biofeedback (Experimental): Real-time visual biofeedback of braking forces during a treadmill run.
  Interventions: Device: Real-time visual biofeedback during treadmill running

INTERVENTIONS:
Device: Real-time visual biofeedback during treadmill running — Real-time biofeedback of braking forces during running

SUMMARY:
The proposed research study aims to investigate whether a gait modification training program to decrease peak braking forces during the stance phase of running will result in a reduction in impact loading and the incidence of running-related injuries among recreational distance runners.

ELIGIBILITY:
Inclusion Criteria:

* Ability to commit to a 15-week half-marathon training program
* Have been running for at least 3 months prior to study commencement
* Have participated in 2 or less half-marathons previously
* Ability to run on a treadmill unaided
* Ability to travel to testing facility for running analysis pre- and post-training program as well as for gait retraining sessions
* Ability to understand written and spoken English
* Meet the screening requirements (display less than -0.27BW mean peak braking force at baseline/screening assessment)

Exclusion Criteria:

* Any lower extremity pathology in the previous 3 months or currently have pain in their lower back or lower extremities while running
* Have undergone hip, knee, or ankle joint surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Hunt, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Fortius Sport & Health, Burnaby, British Columbia, Canada

REFERENCES:
- [Derived] Napier C, MacLean CL, Maurer J, Taunton JE, Hunt MA. Real-Time Biofeedback of Performance to Reduce Braking Forces Associated With Running-Related Injury: An Exploratory Study. J Orthop Sports Phys Ther. 2019 Mar;49(3):136-144. doi: 10.2519/jospt.2019.8587. Epub 2018 Dec 7. PMID 30526232

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real Time Biofeedback
Started | 16
Completed | 12
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Real Time Biofeedback
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 12
Peak Braking Force [Mean (Standard Deviation); unit: Body Weight] | 0.28 (0.04)
Step Length [Mean (Standard Deviation); unit: m] | 0.91 (0.07)

OUTCOME MEASURES:

1. Primary Outcome: Peak Braking Force
Description: The peak horizontal force applied in the posterior direction during the stance phase of running
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: Body Weight
Arm/Group | Real Time Biofeedback
Number analyzed (Participants) | 12
Body Weight | 0.24 (0.02)
Statistical Analysis 1: Comparison: Real Time Biofeedback; Test type: Superiority; p = 0.001, ANOVA

2. Secondary Outcome: Average Vertical Loading Rate
Description: The average vertical loading rate during stance phase
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: Body Weight/second
Arm/Group | Real Time Biofeedback
Number analyzed (Participants) | 12
Body Weight/second | 36.05 (7.5)

3. Secondary Outcome: Step Length
Description: The average step length
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Real Time Biofeedback
Number analyzed (Participants) | 12
m | 0.85 (0.05)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 15-week period over the course of the running training program.
Description: Adverse events were assessed using open-ended questions in the weekly questionnaire. For the purpose of analysis, adverse events were defined as new pain or discomfort lasting longer than 2 weeks in duration or requiring treatment.
Arm/Group | Real Time Biofeedback
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03302975/Prot_SAP_000.pdf